CLINICAL TRIAL: NCT04919941
Title: A Pilot Study of A Guide to Conservative Care
Brief Title: A Guide to Conservative Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, Susan Wong, Assistant Professor, School of Medicine: Nephrology, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: STUDY00010555; Pilot/Exploratory Grant (Other Grant/Funding Number: National Palliative Care Research Center)
Record Dates: First submitted 2021-05-28; First posted 2021-06-09 (Actual); Last update posted 2022-06-24 (Actual); Status verified 2021-06

CONDITIONS: End Stage Renal Disease; Decision Aid; Patient Engagement; Dialysis; End-of-life Care
Keywords: conservative care
MeSH Terms: conditions — Kidney Failure, Chronic; Patient Participation

STUDY DESIGN:
Intervention Model Description: Test feasibility and acceptability of a patient decision aid
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Decision aid (Experimental): The intervention is receipt of a patient decision aid on conservative care, entitled A Guide to Conservative Care. This is 12-page printed handout that provides an overview of conservative care. Participants assigned to the intervention group are mailed a copy of the Guide after their initial baseline visit (T1). Participants keep the Guide throughout the duration of the study.
  Interventions: Other: A Guide to Conservative Care
- Control (No Intervention): Did not receive the decision aid.

INTERVENTIONS:
Other: A Guide to Conservative Care — The intervention is receipt of a patient decision aid on conservative care, entitled A Guide to Conservative Care. This is 12-page printed handout that provides an overview of conservative care. Participants assigned to the intervention group are mailed a copy of the Guide after their initial baseline visit (T1). Participants keep the Guide throughout the duration of the study.
  Arms: Decision aid

SUMMARY:
This is a randomized pilot study to test the feasibility and acceptability of a patient decision aid on conservative care among older patients with advanced CKD and their close persons.

DETAILED DESCRIPTION:
Conservative care is an important therapeutic option for patients with advanced chronic kidney disease (CKD) who do not wish to pursue maintenance dialysis. However, most patient educational materials on treatment options for advanced CKD do not include information.

This study is a randomized pilot study to test the acceptability and feasibility of a novel patient decision aid on conservative care, entitled A Guide to Conservative Care, among older patients with advanced CKD and their close persons. The investigators hypothesize that the Guide will be feasible and acceptable to patients and families as reflected in greater discussion of conservative care with health care providers following receipt of the Guide as compared with usual care.

The study will enroll 92 patients aged 75 years and older with advanced CKD and up to 92 of their close persons from University of Washington Medicine and Veterans Affairs Puget Sound Health Care System. Enrolled patients are invited but not required to nominate a close person (defined as a person who assists the patient with his/her advanced CKD) to also participate in the study. Patients and their close persons will be randomized together in a 1:1 fashion to receive either the Guide (i.e. intervention) or usual care (i.e. control). Data from participants will be collected at the time of enrollment, 2-week follow-up and 3-month follow-up.

As a reflection of acceptability and feasibility, the primary outcome measure is difference in rates of discussion of conservative care with a healthcare provider at 3-month follow-up. Increased motivation for patients to discuss of conservative care with their health care providers would reflect that the Guide is acceptable to patients and can be feasibly incorporated by them into their care planning. The investigators will also collect completion and attrition rates at the second and third study visits as additional measures of acceptability and feasibility. Furthermore, the investigators will collect feedback on the Guide and experiences with using the Guide from participants who received the Guide using qualitative interviews at 2-week and 3-month follow-up. The investigators will also explore treatment goals and preferences for advanced CKD using standardized surveys at each study visit.

The investigators will use the information gathered during the study towards further refining the Guide so that it will be ready for distribution at participating study sites and future testing in broader patient populations.

ELIGIBILITY:
Inclusion Criteria:

* Patients

  * Adults aged ≥75 years
  * Diagnosis of advanced CKD as defined as having at least 2 outpatient measures of eGFR <25 ml/min/1.73m2 separated by >90 days in the prior year and with at least 1 of these measures of eGFR <20 ml/min/1.73m2
  * Must be english-speaking
* Close persons

  * Adults aged ≥18 years
  * Must assist patient with their kidney disease care
  * Must be English-speaking

Exclusion Criteria:

-Patients and Close Person

• Unable to provide informed consent

Min Age: 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 92 (Actual)
Dates: Start 2020-08-31 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
Questionnaire on patient-provider discussions of conservative care . | 3 months
  Using a questionnaire, patients will be asked whether they had discussed conservative care with any of their healthcare providers prior to T1 and by T3. Possible responses are "yes", "no" or "unsure." Greater motivation to discuss conservative care with their care providers at T3 after would indicate that the Guide is acceptable to patients and can be feasibly incorporated by them into their care planning.
Attrition | 3 months
  The proportion of participants in each study arm who withdraw from the study and the reasons why at T2 and T3. Study withdrawal would indicate that the Guide and/or study is unacceptable or burdensome to the participant.

SECONDARY OUTCOMES:
Treatment Preference | 3 months
  Preference for dialysis or conservative care will be assessed using the Decision Conflict Scale (DCS) at each study visit. The DCS is a16-item survey to assess their level of difficulty in choosing between dialysis vs. conservative care based on uncertainty, values clarity and feeling informed and supported in decision-making. Each item is rated from 0-4 (higher scores indicating greater conflict). For close persons, their preference for dialysis or conservative care for the patient will also be assessed using the Decision Conflict Scale at each study visit.
Treatment Goals | 3 months
  For each patient at each study visit, patients about their preference for either extending life, preserving comfort or unsure using a validated survey question. Close persons will also be asked the same question about what they perceive the patients' healthcare goals are at each study visit.
Guide Questionnaire | 2 weeks
  For participants randomized to receive the intervention, at T2, they will complete a survey inquiring whether they reviewed the Guide, the time it took to review the Guide and whether they had made any notes in the Guide.
Guide Interview | 3 months
  For participants randomized to receive the intervention, at T2 and T3, they will complete a qualitative interview inquiring their likes/dislikes about the Guide, what they found useful/not useful about the Guide, what they found difficult about the Guide, suggestions to improve the Guide, and whether the Guide helped to support discussions about conservative care with others and their healthcare providers.

CONTACTS AND LOCATIONS:
Overall Officials: Susan P Wong, MD, Principal Investigator — University of Washington
Locations (2):
- United States (2):
  - VA Puget Sound Health Care System, Seattle, Washington
  - University of Washington Medicine, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
All de-identified individual participant data collected and study protocols will be shared immediately following publication and ending 5 years following article publication with researchers who provide a written request and sound research proposal. Interested researchers can contact the principal investigator directly.
Supporting Information: Study Protocol
Time Frame: Immediately following publication and through 5 years after article publication
Access Criteria: Written request and sound research plan.

REFERENCES:
- [Derived] Wong SPY, Oestreich T, Prince DK, Curtis JR. A Patient Decision Aid About Conservative Kidney Management in Advanced Kidney Disease: A Randomized Pilot Trial. Am J Kidney Dis. 2023 Aug;82(2):179-188. doi: 10.1053/j.ajkd.2022.12.007. Epub 2023 Feb 4. PMID 36740038

DOCUMENTS (1):
  • Study Protocol (2021-02-23): https://cdn.clinicaltrials.gov/large-docs/41/NCT04919941/Prot_000.pdf